CLINICAL TRIAL: NCT02707445
Title: Prospective Multi-center Registry of Genotyping Related Clopidogrel in Percutaneous Coronary Intervention Patients
Brief Title: Genotyping Influences Outcome of Coronary Artery Stenting
Acronym: GENIUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Do-sun Lim, MD, PhD, Korea University Anam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KUMC-GENIUS
Record Dates: First submitted 2016-02-23; First posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Myocardial Ischemia; CLOPIDOGREL, POOR METABOLISM of (Disorder)
MeSH Terms: conditions — Myocardial Ischemia | interventions — Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GENIUS (Experimental): All comer patients who had undergone percutaneous coronary intervention with administration of conventional dual anti-platelet treatment (aspirin 100mg and clopidogrel 75mg daily) for minimum 3 months
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — Administration of conventional dual anti-platelet treatment (aspirin 100mg and clopidogrel 75mg daily) for minimum 3 months after percutaneous coronary intervention
  Other Names: clopidogrel hydrogen sulfate 97.875mg (75mg as clopidogrel)

SUMMARY:
This study evaluated epidemiology and clinical outcome of clopidogrel related various genotyping in Korean patients who had undergone percutaneous coronary intervention as a all comer registry form.

DETAILED DESCRIPTION:
This study evaluates the relationship between clopidogrel related various genotyping, epidemiology and clinical outcome of patient who had undergone percutaneous coronary intervention. Clopidogrel resistance was measured with VerifyNow, which is a device that can monitor platelet inhibition of clopidogrel. Genes which are known to be related with clopidogrel resistance were evaluated; (1-3) CYP 2C19 *2, *3, *17, (4) PON1 Q192R, (5) ABCB1 3435C->T, (6) P2Y12, (7) CYP 2C9 *3.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Older than 20 years
* All percutaneous coronary intervention patients within 1 month

Exclusion Criteria:

* Pregnancy
* Life expectancy below 1 year
* Known aspirin or clopidogrel allergy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Actual)
Dates: Start 2011-09; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Myocardial infarction and Death | 1 year after index procedure

SECONDARY OUTCOMES:
Any death | 1 year after index procedure
Cardiac death | 1 year after index procedure
Myocardial infarction | 1 year after index procedure
Stent thrombosis (acute, late, very late) | 1 year after index procedure
Target lesion revascularization | 1 year after index procedure
  Revascularization of in-stent restenosis which developed in previously implanted stent on index procedure
Stroke | 1 year after index procedure
  Ischemic or hemorrhagic cerebral infarction diagnosed by brain MRI which developed within 1 year after index procedure
Bleeding complication | During index procedure
PRU | Within index procedure
  Value which is measured with VerifyNow that can monitor platelet inhibition of clopidogrel
ARU | Within index procedure
  Value which is measured with VerifyNow that can monitor platelet inhibition of aspirin

CONTACTS AND LOCATIONS:
Overall Officials: Do-sun Lim, MD, PhD, Principal Investigator — Cardiovascular center, Korea University Anam Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fuster V, Stein B, Ambrose JA, Badimon L, Badimon JJ, Chesebro JH. Atherosclerotic plaque rupture and thrombosis. Evolving concepts. Circulation. 1990 Sep;82(3 Suppl):II47-59. PMID 2203564
- [Result] Storey RF, Newby LJ, Heptinstall S. Effects of P2Y(1) and P2Y(12) receptor antagonists on platelet aggregation induced by different agonists in human whole blood. Platelets. 2001 Nov;12(7):443-7. doi: 10.1080/09537100120085450. PMID 11674863
- [Result] Angiolillo DJ, Fernandez-Ortiz A, Bernardo E, Alfonso F, Macaya C, Bass TA, Costa MA. Variability in individual responsiveness to clopidogrel: clinical implications, management, and future perspectives. J Am Coll Cardiol. 2007 Apr 10;49(14):1505-16. doi: 10.1016/j.jacc.2006.11.044. Epub 2007 Mar 26. PMID 17418288
- [Result] Task Force on Myocardial Revascularization of the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS); European Association for Percutaneous Cardiovascular Interventions (EAPCI); Wijns W, Kolh P, Danchin N, Di Mario C, Falk V, Folliguet T, Garg S, Huber K, James S, Knuuti J, Lopez-Sendon J, Marco J, Menicanti L, Ostojic M, Piepoli MF, Pirlet C, Pomar JL, Reifart N, Ribichini FL, Schalij MJ, Sergeant P, Serruys PW, Silber S, Sousa Uva M, Taggart D. Guidelines on myocardial revascularization. Eur Heart J. 2010 Oct;31(20):2501-55. doi: 10.1093/eurheartj/ehq277. Epub 2010 Aug 29. No abstract available. PMID 20802248
- [Result] Wright RS, Anderson JL, Adams CD, Bridges CR, Casey DE Jr, Ettinger SM, Fesmire FM, Ganiats TG, Jneid H, Lincoff AM, Peterson ED, Philippides GJ, Theroux P, Wenger NK, Zidar JP, Anderson JL, Adams CD, Antman EM, Bridges CR, Califf RM, Casey DE Jr, Chavey WE 2nd, Fesmire FM, Hochman JS, Levin TN, Lincoff AM, Peterson ED, Theroux P, Wenger NK, Wright RS. 2011 ACCF/AHA focused update of the Guidelines for the Management of Patients with Unstable Angina/Non-ST-Elevation Myocardial Infarction (updating the 2007 guideline): a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines developed in collaboration with the American College of Emergency Physicians, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. J Am Coll Cardiol. 2011 May 10;57(19):1920-59. doi: 10.1016/j.jacc.2011.02.009. Epub 2011 Mar 28. No abstract available. PMID 21450428
- [Result] Schomig A. Ticagrelor--is there need for a new player in the antiplatelet-therapy field? N Engl J Med. 2009 Sep 10;361(11):1108-11. doi: 10.1056/NEJMe0906549. Epub 2009 Aug 30. No abstract available. PMID 19717845
- [Result] Simon T, Verstuyft C, Mary-Krause M, Quteineh L, Drouet E, Meneveau N, Steg PG, Ferrieres J, Danchin N, Becquemont L; French Registry of Acute ST-Elevation and Non-ST-Elevation Myocardial Infarction (FAST-MI) Investigators. Genetic determinants of response to clopidogrel and cardiovascular events. N Engl J Med. 2009 Jan 22;360(4):363-75. doi: 10.1056/NEJMoa0808227. Epub 2008 Dec 22. PMID 19106083
- [Result] Mega JL, Simon T, Collet JP, Anderson JL, Antman EM, Bliden K, Cannon CP, Danchin N, Giusti B, Gurbel P, Horne BD, Hulot JS, Kastrati A, Montalescot G, Neumann FJ, Shen L, Sibbing D, Steg PG, Trenk D, Wiviott SD, Sabatine MS. Reduced-function CYP2C19 genotype and risk of adverse clinical outcomes among patients treated with clopidogrel predominantly for PCI: a meta-analysis. JAMA. 2010 Oct 27;304(16):1821-30. doi: 10.1001/jama.2010.1543. PMID 20978260
- [Result] Bouman HJ, Schomig E, van Werkum JW, Velder J, Hackeng CM, Hirschhauser C, Waldmann C, Schmalz HG, ten Berg JM, Taubert D. Paraoxonase-1 is a major determinant of clopidogrel efficacy. Nat Med. 2011 Jan;17(1):110-6. doi: 10.1038/nm.2281. Epub 2010 Dec 19. PMID 21170047
- [Result] Gladding P, White H, Voss J, Ormiston J, Stewart J, Ruygrok P, Bvaldivia B, Baak R, White C, Webster M. Pharmacogenetic testing for clopidogrel using the rapid INFINITI analyzer: a dose-escalation study. JACC Cardiovasc Interv. 2009 Nov;2(11):1095-101. doi: 10.1016/j.jcin.2009.08.018. PMID 19926050
- [Result] Fontana P, Dupont A, Gandrille S, Bachelot-Loza C, Reny JL, Aiach M, Gaussem P. Adenosine diphosphate-induced platelet aggregation is associated with P2Y12 gene sequence variations in healthy subjects. Circulation. 2003 Aug 26;108(8):989-95. doi: 10.1161/01.CIR.0000085073.69189.88. Epub 2003 Aug 11. PMID 12912815
- [Result] Luo HR, Poland RE, Lin KM, Wan YJ. Genetic polymorphism of cytochrome P450 2C19 in Mexican Americans: a cross-ethnic comparative study. Clin Pharmacol Ther. 2006 Jul;80(1):33-40. doi: 10.1016/j.clpt.2006.03.003. Epub 2006 Jun 8. PMID 16815315
- [Result] Trenk D, Hochholzer W, Fromm MF, Chialda LE, Pahl A, Valina CM, Stratz C, Schmiebusch P, Bestehorn HP, Buttner HJ, Neumann FJ. Cytochrome P450 2C19 681G>A polymorphism and high on-clopidogrel platelet reactivity associated with adverse 1-year clinical outcome of elective percutaneous coronary intervention with drug-eluting or bare-metal stents. J Am Coll Cardiol. 2008 May 20;51(20):1925-34. doi: 10.1016/j.jacc.2007.12.056. PMID 18482659
- [Derived] Cha JJ, Joo HJ, Park JH, Hong SJ, Ahn TH, Kim BK, Shin W, Ahn SG, Yoon J, Kim YH, Cho YH, Kang WC, Kim W, Lim YH, Gwon H, Choi W, Lim DS. Impact of genetic variants on major bleeding after percutaneous coronary intervention based on a prospective multicenter registry. Sci Rep. 2021 Jan 19;11(1):1790. doi: 10.1038/s41598-020-80319-9. PMID 33469058